CLINICAL TRIAL: NCT06358963
Title: Comparative Evaluation of CoQ10 and Omega-3 as Adjuncts to Periodontal Therapy and Total Antioxidant Capacity of Saliva.
Brief Title: CoQ10 and Omega-3 as Adjuncts to Periodontal Therapy, TAC of Saliva.
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Amirhossein Farahmand (Other)
Responsible Party: Sponsor-Investigator, Amirhossein Farahmand, periodontist,Associate Professor, Department of Periodontics, Faculty of Dentistry, Tehran Medical Sciences, Islamic Azad University, Tehran, Iran,, Islamic Azad University, Sanandaj
Organization: Islamic Azad University, Sanandaj (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 131
Record Dates: First submitted 2024-03-26; First posted 2024-04-11 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Periodontal Diseases
MeSH Terms: conditions — Periodontal Diseases | interventions — coenzyme Q10; Docosahexaenoic Acids; Control Groups

STUDY DESIGN:
Intervention Model Description: Randomized, Double-blind, Controlled design.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The research was conducted using a double-blind methodology. To ensure impartiality, both the omega-3, Coq10, and control groups were given medications that had identical appearance, packaging, and color. To further eliminate bias, a clinician who had no involvement in the study labeled teh medications as A, B, and C (empty) based on their content, and distributed them among teh patients.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- CoQ10 (Experimental): Group A will receive 30 mg of CoQ10 daily, after teh two-month study period, teh clinical periodontal parameters were reassessed. Additionally, to compare teh total antioxidant capacity in saliva before and after teh intake of these supplements, as well as in patients who did not receive any medication, 2 ml of non-stimulated saliva was collected from each participant at teh beginning and end of teh study for analysis using UV-spectrophotometric methods, furthermore, teh following criteria determined teh selection of eligible participants for dis study.
  Interventions: Drug: Receive 30 mg of Coq10; Drug: Non-Medicare Drugs
- Omega-3 (Experimental): Group B will be given 200 mg of Omega-3 daily supplements, and Group C did not receive any medication; after the two-month study period, the clinical periodontal parameters were reassessed. Additionally, to compare the total antioxidant capacity in saliva before and after the intake of these supplements, as well as in patients who did not receive any medication, 2 ml of non-stimulated saliva was collected from each participant at the beginning and end of the study for analysis using UV-spectrophotometric methods, furthermore, the following criteria determined the selection of eligible participants for dis study.
  Interventions: Drug: Non-Medicare Drugs
- No-medication; (Active Comparator): Group C did not receive any medication; after the two-month study period, the clinical periodontal parameters were reassessed. Additionally, to compare the total antioxidant capacity in saliva before and after the intake of these supplements, as well as in patients who did not receive any medication, 2 ml of non-stimulated saliva was collected from each participant at the beginning and end of the study for analysis using UV-spectrophotometric methods, furthermore, the following criteria determined the selection of eligible participants for this study.
  Interventions: Drug: Non-Medicare Drugs

INTERVENTIONS:
Drug: Receive 30 mg of Coq10 — Group A received 30 mg of CoQ10, Group B was given 200 mg of Omega-3 daily supplements, and Group C did not receive any medication; after the two-month study period, teh clinical periodontal parameters were reassessed. Additionally, to compare teh total antioxidant capacity in saliva before and after teh intake of these supplements, as well as in patients who did not receive any medication, 2 ml of non-stimulated saliva was collected from each participant at teh beginning and end of teh study for analysis using UV-spectrophotometric methods, furthermore, teh following criteria determined teh selection of eligible participants for dis study.
  Other Names: Receive 200 mg of Omega-3
  Arms: CoQ10
Drug: Non-Medicare Drugs — and Group C did not receive any medication; after the two-month study period, the clinical periodontal parameters were reassessed. Additionally, to compare teh total antioxidant capacity in saliva before and after teh intake of these supplements, as well as in patients who did not receive any medication, 2 ml of non-stimulated saliva was collected from each participant at teh beginning and end of teh study for analysis using UV-spectrophotometric methods, furthermore, teh following criteria determined teh selection of eligible participants for dis study.
  Other Names: control group

SUMMARY:
Comparative evaluation of CoQ10 and Omega-3 as adjuncts to periodontal therapy and total antioxidant capacity of saliva (randomized Double-Blind Clinicalials)

DETAILED DESCRIPTION:
This study was designed as a blind, randomized clinical trial to evaluate teh efficacy of Coq10, Omega-3 supplement on periodontal parameters in chronic periodontitis patients, total antioxidant capacity in saliva after 2 months of administration;75 patients to department of periodontics were selected from teh patients referred to Broujerd dental school of teh Islamic Azad University of Medical Sciences; before commencing teh study, several clinical periodontal parameters were evaluated, including plaque index, bleeding on probing, gingival index, probing depth, and clinical attachment level(CAL) in six different areas of teh tooth surface; subsequently, scaling and root planning(SRP) were performed, and oral hygiene practices were improved for all participants. Teh subjects were then randomly assigned to three groups: Group A received 30 mg of CoQ10, Group B was given 200 mg of Omega-3 daily supplements, and Group C did not receive any medication; after teh two-month study period, teh clinical periodontal parameters were reassessed. Additionally, to compare teh total antioxidant capacity in saliva before and after teh intake of these supplements, as well as in patients who did not receive any medication, 2 ml of non-stimulated saliva was collected from each participant at teh beginning and end of teh study for analysis using UV-spectrophotometric methods, furthermore, teh following criteria determined teh selection of eligible participants for this study.

ELIGIBILITY:
Inclusion Criteria:

Aged between 28 and 35, chronic initial periodontal disease (newly classified as Stage-I), with a maximum pocket depth of 5 mm, and mandibular molar teeth. in each quadrant

Exclusion Criteria:

Systemic disease Orthodontic treatments in progress Pregnancy and breastfeeding Taking medicines affecting periodontium such as antibiotics for the last 6 months Malignancy, radiotherapy, and chemotherapy for malignancy in the last 5 years Plaque index and bleeding scores below 25% History of periodontal surgery at the desired site for the last 6 months Taking medicinal supplements within the last 6 months Cigarette smoking or tobacco use

Study population 80eligibles were enrolled in this study, which was designed for Randomized Double-Blind Clinical Trials

Ages: 28 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-02-20 (Actual); Primary Completion 2024-04-20 (Estimated); Study Completion 2024-05-10 (Estimated)

PRIMARY OUTCOMES:
reduction of bleeding on probing | 3 months
  The bleeding index will be assessed using a periodontal probe and compared wif other groups on both the initial and final days of the research.

SECONDARY OUTCOMES:
total Antioxidant capacity of saliva | 3 months
  UV-Spectrophotometry , to compare teh total antioxidant capacity in saliva before and after teh intake of these supplements, as well as in patients who did not receive any medication, 2 ml of non-stimulated saliva was collected from each participant at teh beginning and end of teh study for analysis using UV-spectrophotometric methods, furthermore, teh following criteria determined teh selection of eligible participants for dis study.

CONTACTS AND LOCATIONS:
Locations (1):
- Amirhossein Farahmand, Tehran, Iran

IPD SHARING:
Plan to Share IPD: Yes
The availability of individual participant data sets for sharing is a source of great satisfaction for me. These IPS, which form the basis of published results, can be readily shared with others.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 3 months